CLINICAL TRIAL: NCT02166606
Title: INGEVITY™ Observational Trial: Assessment of Routine Experience and Magnet Resonance Imaging (MRI) Usage With a New Lead for Bradycardia Pacing
Brief Title: INGEVITY™ Observational Trial
Acronym: GENTLE
Status: Completed | Type: Observational
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: GENTLE-1013
Record Dates: First submitted 2014-04-11; First posted 2014-06-18 (Estimated); Results first posted 2019-08-20 (Actual); Last update posted 2021-03-30 (Actual); Status verified 2019-08

CONDITIONS: Bradycardia
MeSH Terms: conditions — Bradycardia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Pacemaker/Lead implant: All enrolled subjects will receive an ImageReady Magnet Resonant (MR) Conditional Pacing System and the treatment assignment will be based on an "all-comers" consecutive basis.
  Interventions: Device: ImageReady MR Conditional Pacing System Implant

INTERVENTIONS:
Device: ImageReady MR Conditional Pacing System Implant — Implant according to standard-of-care. No study-specific interventions in that registry.

SUMMARY:
The objectives of this registry are to

1. Collect clinical data on Boston Scientific's ImageReady MR Conditional Pacing Systems involving the INGEVITY lead based on observations / events
2. Gather data on actual number of MRI scans performed in the patient cohort implanted with an ImageReady system including information about scanned body parts.
3. Collect physician feedback on lead handling with the INGEVITY lead

in a real-life, market-released standard of care environment using devices on intended purpose and which are authorized to bear the CE (Communauté Européenne) marking / are approved for use in the applicable area of participating centers. No additional invasive or other burdensome examinations are to be carried out other than the ones conducted by the centers per their general standard of care.

ELIGIBILITY:
Inclusion Criteria:

* Subject is willing and capable of providing informed consent and to give approval to collect / store / process personal health information by the sponsor
* Subject is scheduled for, or implanted with, a clinically indicated BSC ImageReady system according to current and locally applicable implant guidelines such as published by European Society of Cardiology (ESC) / American Heart Association (AHA) / American College of Cardiology (ACC) / Hearth Rhythm Society (HRS)
* Subject is geographically stable to be available for follow up at an approved registry center during the whole registry duration
* Subject is age 18 or above, or of legal age to give informed consent specific to state and national law

Exclusion Criteria:

* Existing contraindications for a BSC ImageReady system as mentioned in the applicable reference guides of the implanted system components including a known or suspected sensitivity to dexamethasone acetate (DXA)
* Implanted pacing system is not ImageReady, i.e. any system components other than BSC INGEVITY MRI Conditional leads (or their market released successors), BSC INGENIO MRI family pacemaker models and their accessories (or their market released successors) intended to have MR Conditional status, including pre-existing abandoned leads of any kind still implanted and which will not be removed during the implant or re-implant procedure or plugged lead ports
* Any existing conditions per local standard of care preventing the subject from undergoing an MRI procedure including implanted active or inactive medical devices / material, not considered MR Conditional
* Subject is enrolled in any other concurrent study with the exception of local mandatory governmental registries and studies/registries that are not in conflict and do not affect the following:

  1. GENTLE registry outcome (i.e. involve different implantable system components than required for participation in GENTLE or would affect ability to undergo MRI procedures);
  2. Conduct of the GENTLE Registry per Good Clinical Practice (GCP)/ ISO (International Organization of Harmonization) 14155:2011/ local regulations as applicable
* Subject is a woman of childbearing potential who is, or might be, pregnant at the time of registry enrollment or plans to become pregnant during the course of the registry (based on physician's assessment)
* Estimated life expectancy of less than twelve months per physician discretion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The subjects will be coming from the general patient population of the participating centers who are indicated for implantation of a BSC (Boston Scientific) ImageReady Pacing System (pulse generator [PG] & leads) and who are fulfilling all inclusion criteria and none of the exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 1184 (Actual)
Dates: Start 2014-04 (Actual); Primary Completion 2016-06 (Actual); Study Completion 2016-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Gras, MD, Principal Investigator — Nouvelles Cliniques Nantaises Cardiologie / Médecins du pôle - Unité de Soins et de Cardiologie Interventionnelle 4 rue Eric Tabarly 44277 Nantes cedex 2 France; John doe, MD, Principal Investigator
Locations (60):
- Austria (2):
  - Medizinische Universitat Graz, Graz
  - AKh - Allgemeines Krankenhaus der Stadt Linz GmbH, Linz
- Belgium (4):
  - Ziekenhaus Oost Limburg, Genk
  - Grand Hopital De Charleroi, Gilly
  - Jessa Hospital, Hasselt
  - UCL de Mont Godinne, Yvoir
- France (15):
  - Clinique Rhone Durance, Avignon
  - Hopital Prive Saint Martin, Caen
  - Centre Hospitalier du Contentin, Cherbourg
  - Centre Hospitalier de Marne La Vallee, Jossigny
  - Hopital Saint Philibert, Lomme
  - Hopital Prive Jacques Cartier, Massy
  - Clinique Les Fontaines, Melun
  - Centre Hospitalier de Moulins, Moulins
  - Le Confluent - Nouvelles Cliniques Nantaises, Nantes
  - Hopital Regional Orleans La Source, Orléans
  - Groupement Hospitalier Pitie Salpetriere, Paris
  - Centre Hospitalier Universitaire de Poitiers, Poitiers
  - Centre Hospitalier de Saintonge, Saintes
  - Clinique Saint Gatien, Tours
  - Centre Hospitalier Bretagne Atlantique, Vannes
- Germany (7):
  - Charite, Universitatsmedizin Berlin, Campus Benjamin Franklin, Klinik fur Kardiologie und Pulmologie, Berlin
  - Unfallkrankenhaus Berlin, Klinik fur Innere Medizin, Berlin
  - Immanuel Klinikum Bernau/Herzzentrum Brandenburg, Bernau
  - Universitatsklinikum Dusseldorf, Klinik fur Kardiovaskulare Chrirurgie, Düsseldorf
  - Cardioangiologisches Centre Bethanien, Frankfurt
  - Herz- und Gefäßzentrum am Krankenhaus Neu-Bethlehem, Göttingen
  - St. Marienkrankenhaus Siegen, Siegen
- Ireland (2):
  - University Hospital Galway, Galway
  - Bon Secours Hospital, Tralee
- Italy (7):
  - Fondazione Poliambulanza, Brescia
  - Ospedale Annunziata, Cosenza
  - Ospedale Spaziani Frosinone, Frosinone
  - Ospedale Guzzardi di Vittoria, Ragusa
  - Policlinico Casilino, Roma
  - Azienda ULSS 9 Treviso, Treviso
  - Ospedale Borgo Trento, Verona
- Akershus Universitetssykehus HF, Lorenskog, Norway
- Portugal (5):
  - Hospital Professor Doutor Fernando Fonseca, EPE, Amadora
  - Centro Hospitalar do Alto Ave, EPE, Guimarães
  - CHLO, EPE, Hospital S. Francisco Xavier, Lisbon
  - CHLN, EPE Hospital de Santa Maria, Lisbon
  - Hospital dos SAMS, Lisbon
- South Korea (5):
  - Seoul National University Bundang Hospital, Gyeonggi-do
  - Korea University Anam Hospital, Seoul
  - Seoul National University Hospital, Seoul
  - Yonsei University Severance Hospital, Seoul
  - Samsung Medical Center, Seoul
- Spain (8):
  - Hospital Clinic de Barcelona, Barcelona
  - Hospital Universitario Infanta Leonor, Madrid
  - Hospital Universitario Ramon y Cajal, Madrid
  - Hospital Puerta de Hierro, Majadahonda
  - Hospital de Merida, Mérida
  - Hospital Universitario Nuestra Senora de Candelaria, Santa Cruz de Tenerife
  - Hospital Clinico Universitario Valladolid, Valladolid
  - Hospital Virgen de la Concha, Zamora
- Sweden (2):
  - Skanes Universitetssjukhus, Lund
  - St Gorans Sjukhus, Stockholm
- Universitatsspital Basel, Basel, Switzerland
- Morriston Hospital, Swansea, United Kingdom

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrollment in the study began on 02 April 2014. The enrollment completion for the GENTLE study was communicated to the participating sites on 26 February 2016. However, additional subjects were enrolled after this date and the last subject signed consent on 08 March 2016. The last subject last visit was on 07 June 2016.
Pre-assignment Details: 1184 subjects signed the informed consent (IC). 4 subjects signed the IC only after the end of enrollment. 1180 subjects signed IC before the end of enrollment and are considered 'actively enrolled'. 1174 subjects met all eligibility criteria and were thus considered 'consent eligible' and were considered for the baseline.
Groups:
- Pacemaker/Lead Implant: All enrolled subjects received an ImageReady Magnet Resonant (MR) Conditional Pacing System according to standard-of-care. No study-specific interventions were performed in the registry. The treatment assignment was based on an "all-comers" consecutive basis.
Period: Overall Study
Arm/Group | Pacemaker/Lead Implant
Started | 1184
Actively Enrolled | 1180
Consent Eligible | 1174
Completed | 1106
Not Completed | 78
Not completed — Adverse Event | 3
Not completed — Death | 31
Not completed — Protocol Violation | 7
Not completed — Lost to Follow-up | 30
Not completed — Withdrawal by Subject | 1
Not completed — Physician Decision | 1
Not completed — Device upgrade | 1
Not completed — Enrolled after End of Enrollment | 4

BASELINE CHARACTERISTICS:
Groups:
- Pacemaker/Lead Implant: All enrolled subjects will receive an ImageReady Magnet Resonant (MR) Conditional Pacing System and the treatment assignment will be based on an "all-comers" consecutive basis.
  ImageReady MR Conditional Pacing System Implant: Implant according to standard-of-care.
  No study-specific interventions in that registry.
Arm/Group | Pacemaker/Lead Implant
Number analyzed (Participants) | 1174
Age, Continuous [Mean (Standard Deviation); unit: years] | 74.8 (10.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 413
  Male | 761
Region of Enrollment [Number; unit: participants]
  United Kingdom | 4
  Portugal | 75
  Switzerland | 8
  Spain | 170
  Austria | 38
  South Korea | 20
  Sweden | 13
  Belgium | 84
  Norway | 16
  Ireland | 45
  Italy | 208
  France | 372
  Germany | 121
Primary Brady Indication [Number; unit: participants]
  None | 0
  Sinus bradycardia | 92
  Sinus node dysfunction | 249
  Sinus arrest | 51
  Chronotropic incompetence | 17
  1st degree AV block | 33
  2nd degree AV block | 247
  3rd degree AV block | 293
  Other | 192

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Leads Free From Complication
Description: Lead-related complication-free rate from lead implant through the three month follow-up, based on complications that are related to the INGEVITY Lead.
Time Frame: 91 calendar days post-implant
Measure: Mean (95% Confidence Interval); unit: percentage of leads complication-free
Groups:
- Pacemaker/Lead Implant: All enrolled subjects successfully implanted with a complete ImageReady™ System.
Arm/Group | Pacemaker/Lead Implant
Number analyzed (Participants) | 1174
percentage of leads complication-free | 97.3 [96.2 to 98.1]

2. Other Pre Specified Outcome: MRI Procedures Through 12 Months Post-Implant
Description: The percentage of subjects who underwent an MRI scan through 12 months post-implant.
Time Frame: 365 calendar days post implant
Measure: Number; unit: Percentage of subjects with MRI Scan
Arm/Group | Pacemaker/Lead Implant
Number analyzed (Participants) | 1174
Percentage of subjects with MRI Scan | 2.3

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Pacemaker/Lead Implant
All-Cause Mortality (participants affected / at risk) | 31/1174
Serious Adverse Events (participants affected / at risk) | 197/1174
Other Adverse Events (participants affected / at risk) | 0/1174
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pacemaker/Lead Implant (N=1174)
Non-Cardiovascular/General (Gastrointestinal disorders) | 14 — Gastrointestinal
Non-Cardiovascular/General (General disorders) | 13 — Death
Non-Cardiovascular/General (General disorders) | 10 — Cancer
Non-Cardiovascular/General (Respiratory, thoracic and mediastinal disorders) | 10 — Pulmonary
Non-Cardiovascular/General (Injury, poisoning and procedural complications) | 7 — Physical trauma
Non-Cardiovascular/General (Renal and urinary disorders) | 6 — Genitourinary
Non-Cardiovascular/General (Nervous system disorders) | 6 — Neurological
Non-Cardiovascular/General (General disorders) | 6 — Other - Subject condition - Non- cardiovascular
Non-Cardiovascular/General (Musculoskeletal and connective tissue disorders) | 5 — Musculoskeletal
Non-Cardiovascular/General (Renal and urinary disorders) | 5 — Renal
Non-Cardiovascular/General (Endocrine disorders) | 4 — Endocrine
Non-Cardiovascular/General (General disorders) | 4 — Head, eyes, ears, nose, throat
Non-Cardiovascular/General (General disorders) | 3 — Fever
Non-Cardiovascular/General (Gastrointestinal disorders) | 3 — Integumentary
Non-Cardiovascular/General (Infections and infestations) | 3 — Systemic infection
Non-Cardiovascular/General (Blood and lymphatic system disorders) | 2 — Hematological
Non-Cardiovascular/General (General disorders) | 1 — Abnormal laboratory values
Non-Cardiovascular/General (General disorders) | 1 — Adverse reaction - General
Non-Cardiovascular/General (Psychiatric disorders) | 1 — Psychological
Non-Cardiovascular/General (Nervous system disorders) | 1 — Vasovagal reaction
Atrial Tachyarrhythmias (Cardiac disorders) | 12 — Atrial fibrillation
Atrial Tachyarrhythmias (Cardiac disorders) | 8 — Other Supra Ventricular Tachycardia (SVT)
Atrial Tachyarrhythmias (Cardiac disorders) | 6 — Atrial flutter
Related to Ischemia (Cardiac disorders) | 12 — Coronary artery disease
Related to Ischemia (Cardiac disorders) | 3 — Myocardial infarction
Symptoms (Non-Heart Failure Related) (General disorders) | 4 — Dizziness
Symptoms (Non-Heart Failure Related) (Respiratory, thoracic and mediastinal disorders) | 3 — Chest pain - Other
Symptoms (Non-Heart Failure Related) (Cardiac disorders) | 2 — Chest pain - Ischemic
Symptoms (Non-Heart Failure Related) (Respiratory, thoracic and mediastinal disorders) | 2 — Dyspnea
Symptoms (Non-Heart Failure Related) (General disorders) | 1 — Multiple symptoms
Symptoms (Non-Heart Failure Related) (Cardiac disorders) | 1 — Other - Subject condition - Cardiovascular
Symptoms (Non-Heart Failure Related) (General disorders) | 1 — Syncope
Related to Heart Failure (Cardiac disorders) | 7 — Heart failure symptoms - Unspecified
Related to Heart Failure (Cardiac disorders) | 3 — Dyspnea - Heart failure
Related to Heart Failure (Cardiac disorders) | 3 — Other- Heart failure subject condition - Cardiovascular
Related to Heart Failure (Cardiac disorders) | 1 — Hypertension - Heart failure
Related to Blood Pressure (Vascular disorders) | 3 — Hypertension
Related to Blood Pressure (Vascular disorders) | 1 — Cardiogenic shock
Related to Blood Pressure (Vascular disorders) | 1 — Hypotension
Related to Vasculature (Vascular disorders) | 5 — Peripheral vascular disease
Ventricular Tachyarrythmias (Cardiac disorders) | 3 — Ventricular tachycardia
Ventricular Tachyarrythmias (Cardiac disorders) | 1 — Nonsustained ventricular tachycardia
Thromboembolic Events (Blood and lymphatic system disorders) | 2 — Cerebrovascular accident
Thromboembolic Events (Blood and lymphatic system disorders) | 2 — Pulmonary embolism
Other (Unrelated to Procedure/Device) (Infections and infestations) | 1 — Pericarditis - Unrelated to procedure or device
Right Atrium - Brady (Product Issues) | 9 — Dislodgment - No reported signs - RA
Right Atrium - Brady (Product Issues) | 2 — Other - Lead
Right Atrium - Brady (Product Issues) | 1 — Dislodgment - Elevated threshold - RA
Right Atrium - Brady (Product Issues) | 1 — Elevated threshold - RA
Right Atrium - Brady (Product Issues) | 1 — Impedance > 2000 ohms - RA
Right Atrium - Brady (Product Issues) | 1 — Other - Pulse Generator (PG) system
Right Ventricle - Brady (Product Issues) | 6 — Dislodgment - No reported signs - RV
Right Ventricle - Brady (Product Issues) | 2 — Myocardial perforation post-implant - RV
Right Ventricle - Brady (Product Issues) | 2 — Unable to capture - RV
Right Ventricle - Brady (Product Issues) | 1 — Conductor coil fracture - RV
Right Ventricle - Brady (Product Issues) | 1 — Dislodgment - Multiple signs - RV
Right Ventricle - Brady (Product Issues) | 1 — Dislodgment - Unable to capture - RV
Right Ventricle - Brady (Product Issues) | 1 — Elevated threshold - RV
Procedure (Injury, poisoning and procedural complications) | 6 — Pneumothorax
Procedure (Injury, poisoning and procedural complications) | 2 — Hemothorax
Procedure (Injury, poisoning and procedural complications) | 1 — Other - Lead - Procedure
Procedure (Injury, poisoning and procedural complications) | 1 — Pericardial effusion
PG System - Procedure (Injury, poisoning and procedural complications) | 2 — Hematoma - Pocket (≤ 30 days post-implant)
PG System - Procedure (Injury, poisoning and procedural complications) | 1 — Other - PG system - Procedure
PG system - Procedure (Injury, poisoning and procedural complications) | 1 — Post-surgical pocket hemorrhage
Device Deficiency (Product Issues) | 3 — Device Deficiency
Atrial Tachyarrhythmias (Product Issues) | 2 — Other SVT (e.g. AVRT, AVNRT, EAT)
PG System - Subject (Infections and infestations) | 1 — Infection (> 30 days post-implant)
PG System - Therapy (Product Issues) | 1 — Pacemaker-mediated tachycardia
Ventricular Tachyarrythmias (Cardiac disorders) | 1 — Torsades des pointes

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Consultant (PI) acknowledges and agrees that (i) Consultant shall not publish any data, report, white papers or other materials arising out of the Services performed pursuant to this Agreement without the prior written consent of Boston Scientific, and (ii) any such publication shall not include Boston Scientific Confidential Information except prior written consent of Boston Scientific.